CLINICAL TRIAL: NCT06031857
Title: Comparison of Kinesio Tape and Dry Needling for the Management of Rotator Cuff Tendinopathy: A Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuro Counsel Hospital, Pakistan (Other)
Collaborators: Rawal General and Dental hospital, Islamabad (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 343
Record Dates: First submitted 2023-09-04; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Rotator Cuff Tendinopathy
MeSH Terms: interventions — Athletic Tape; Dry Needling

STUDY DESIGN:
Intervention Model Description: Single blind RCT
Who Masked: Participant
Masking Description: Single blind RCT in which just participants were unaware of intervention they are given
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): . Group A was given kinesio tape.Total six sessions of each intervention were given to each patient at a rate of two sessions per week along with the 10 minutes of interferential therapy and 10 minutes of moist packs to each patient
  Interventions: Other: kinesio tape
- Group B (Active Comparator): . Group A was given dry needling. Total six sessions of each intervention were given to each patient at a rate of two sessions per week along with the 10 minutes of interferential therapy and 10 minutes of moist packs to each patient
  Interventions: Other: Dry needling

INTERVENTIONS:
Other: kinesio tape — kinesio tape was applied over the specific muscle of rotator cuff
  Arms: Group A
Other: Dry needling — dry needling was applied over the affected muscles
  Arms: Group B

SUMMARY:
Its a single blind RCT

DETAILED DESCRIPTION:
Kinesio tape and dry needling were compared for the management of rotator cuff tendinopathy

ELIGIBILITY:
Inclusion Criteria:

* age between 25-50 years old
* Both genders
* Not any comorbidity

Exclusion Criteria:

* Parkinson disease
* DM
* HTN

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2023-08-09 (Actual); Study Completion 2023-08-09 (Actual)

PRIMARY OUTCOMES:
PNS | will be used to assess at baseline after 3 weeks
  Pain numeric Scale consists of 10 scores. 0 means no pain and 10 means worst pain ever
SF-36 | will be used to assess at baseline after 3 weeks
  short form 36 is used to measure the quality of life. lower scores means lower quality of life and ligher score means better quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- The Neurocouncil Clinic, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
have not decided yet